CLINICAL TRIAL: NCT01749683
Title: Myocardial Perfusion Study to Detect Coronary Microvascular Abnormality in Diabetic Patients With Nonfatal Myocardial Infarction
Acronym: GEMyCE 1
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: GEMyCE1
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2016-04

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to use MCE (myocardial contrast/perfusion echocardiography) to study and compare short/long term change of myocardial perfusion abnormality and cardiac outcome in diabetic patients after nonfatal MI (heart attack), who are treated with different glucose control agents.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic and nondiabetic patients will be initially recruited and studied after acute nonfatal MI and revascularization with either PCI or CABG

Exclusion Criteria:

* Patients are excluded if they are older than 70 year old, require mechanical ventilation, are receiving intravenous pressors or hemodynamic support, or if the motion of segments associated with infarct-related artery can not be accurately determined.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic and nondiabetic patients will be initially recruited and studied after acute nonfatal MI and revascularization with either PCI or CABG
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Perfusion abnormalities in nondiabetic and diabetic patients | short term (3 month) and long term (12 month).

SECONDARY OUTCOMES:
The effect of different glycemic control strategies on the reduction of coronary injury in diabetic and non-diabetic subjects | short term (3 month) and long term (12 month)

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States